CLINICAL TRIAL: NCT05520242
Title: Use of Small Animations Movies to Increase Response in a National Health Survey. A Random-ised Controlled Trial. A Study Protocol
Brief Title: Use of Animations Movies to Increase Response in a National Health Survey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region Capital Denmark (Other); North Denmark Region (Other Government); Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10.882
Record Dates: First submitted 2021-01-03; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Response; Non-response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): No animation
- General animation movie (Experimental): Participants randomized to receive the general animation video
  Interventions: Other: Use of small animation movies to increase response in a national health survey
- Men aged 16-24 years (Experimental): Participants randomized to receive the animation targeted men aged 16-24 years
  Interventions: Other: Use of small animation movies to increase response in a national health survey
- Women aged 75 years or older (Experimental): Participants randomized to receive the animation targeted women aged 75 years or older
  Interventions: Other: Use of small animation movies to increase response in a national health survey
- Ethnic minorities (Experimental): Participants randomized to receive the animation targeted ethnic minorities
  Interventions: Other: Use of small animation movies to increase response in a national health survey

INTERVENTIONS:
Other: Use of small animation movies to increase response in a national health survey — Inclusion of animation movies in the invitation cover letter to a national health survey is tested in an embedded randomized controlled trial in the Danish National Health Survey 2021.
  Arms: Ethnic minorities; General animation movie; Men aged 16-24 years; Women aged 75 years or older

SUMMARY:
The aim of this study is to examine the potential for animation movies to improve response rates and sample composition in an embedded randomized controlled trial in the Danish National Health Survey 2021. The overall research question is whether cover letters including an animation movie can perform better than generic letters.

DETAILED DESCRIPTION:
The aim of this study is to examine the potential of animation videos to improve response rates and sample composition in an embedded randomized controlled trial in the Danish National Health Survey 2021 (DNHS-2021). The overall research question is whether digital cover letters including an animation video can perform better than digital letters without animations. The proposition is that such letters should increase the willingness of some sample members to participate by means of increased motivation and reduced complexity, and that this will be reflected in higher response rates. In addition to examining whether it can be advantageous for overall response rates to use cover letters including animation videos, this study also examines the effect of different versions of the animation videos across sample subgroups in order to identify how to best target potential non-respondents in future surveys.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or older and living in Denmark at January 1th 2021.
* Able to receive an invitation through a secure electronical mail service (Digital Post).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201200 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
The number of invited individuals who respond to the survey | 3 month
  A respond is registered if the invited sample member responds to at least 1 question

CONTACTS AND LOCATIONS:
Overall Officials: Anne I Christensen, Principal Investigator — University of Southern Denmark
Locations (1):
- National Institute of Public health, University of Southern Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen AI, Lau CJ, Poulsen HS, Ekholm O. Do animation videos increase participation in national health surveys? A randomised controlled trial. BMC Med Res Methodol. 2023 Aug 14;23(1):184. doi: 10.1186/s12874-023-02005-4. PMID 37580666